CLINICAL TRIAL: NCT06890702
Title: A Prospective Observational Cohort Study of Predictive Biomarkers Related With Ischemic Cerebrovascular Disease
Brief Title: Clinical Evaluation of New Biomarkers for Ischemic Cerebrovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Daishi Tian, Prof., Tongji Hospital
Other Study IDs: TJ-IRB202509068
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke; Ischemic Cerebrovascular Disease
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect samples of urine, fecal, cerebrospinal fluid, blood, plaques, emboli, drainage fluid, bone marrow, lymph nodes, pia mater, dura mater and brain tissue etc.al from patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ischemic cerebrovascular disease: clinical diagnosis with ischemic cerebrovascular disease
  Interventions: Diagnostic Test: biomaker levels
- health control: age- and sex-matched control individuals
  Interventions: Diagnostic Test: biomaker levels

INTERVENTIONS:
Diagnostic Test: biomaker levels — this study will discover and validate novel biomarkers (including urine, feces, cerebrospinal fluid, blood, plaques, emboli, drainage fluid, bone marrow, lymph nodes and brain tissue etc al) of ischemic cerebrovascular disease

SUMMARY:
The goal of this single-center prospective observational study is to identify and evaluate new biomarkers for ischemic cerebrovascular disease (ICVD) to aid in early diagnosis, individualized treatment planning, and prognosis prediction in affected patients. The main questions it aims to answer are:

Can specific biomarkers help in identifying high-risk individuals before disease onset? Can these biomarkers predict disease progression and treatment response? Researchers will compare patients diagnosed with ICVD and healthy controls from a medical check-up center to assess differences in biomarker expression and their clinical significance.

Participants will:

Provide blood, cerebrospinal fluid, urine, and stool samples for biomarker analysis.

Undergo clinical imaging (CT, MRI, PET-CT) and functional assessments. Be followed up at 3, 6, 12, 24, 36, and 48 months for clinical outcomes and biomarker changes.

This study aims to develop a comprehensive biomarker-based prediction model to enhance the diagnosis and management of ischemic cerebrovascular disease.

DETAILED DESCRIPTION:
The detaited information about this trial is described below

1. Quality assurance: The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
2. Data check: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data.
3. Source data verification: Medical records, electronic case report forms, and imaging would be processed by certified neurologists.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic cerebrovascular disease has been proved by clinical symptoms and imaging examinations,including transient ischemic attack, cerebral ischemic stroke, steal syndrome, chronic cerebral hypoperfusion, ect al.
* sex and age-matched healthy individuals

Exclusion Criteria:

* Brain CT or MRI showing cerebral hemorrhage (excluded ischemic stroke with hemorrhage transformation)
* With severe systemic disease, are expected to survive < 3 months
* Patients will not able to provide continuous follow-up information

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic cerebrovascular disease admission to Department of Neurology and Neurosurgery, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology from Janurary 1, 2025 - December 31, 2035
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2035-12-27 (Estimated); Study Completion 2038-01-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 10 years
  Death during the follow-up in every single reason
Stroke of any kind | 10 years
  Brain CT or MRI scans will be used to measure whether there is any kind of stroke, including TIA, ischemic stroke, and hemorrhage

SECONDARY OUTCOMES:
Rehospitalization | 10 years
  The rehospitalized times of any circumstances except for admission to hospital only for examination per year will be used to measure the situation
National Institute of Health stroke scale (NIHSS score) | 10 years
  The minimum value is 0, and maximum value is 42, and higher scores mean a worse outcome.
modified Ranking score (mRS) | 10 years
  The minimum value is 0, and maximum value is 6, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dai-Shi Tian, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology,, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No